CLINICAL TRIAL: NCT04221048
Title: Accuracy of Risk Prediction Scores in Pregnant Women With Congenital Heart Disease.
Brief Title: Accuracy of Risk Prediction Scores in Pregnant Women
Acronym: PREG-GUCH
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0591
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Congenital Heart Disease; Pregnancy
Keywords: Risk score; Maternal complication
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PREG-GUCH: Pregnant women with congenital heart diseases
  Interventions: Other: Retrospective observational

INTERVENTIONS:
Other: Retrospective observational — Pregnancy scores will be based on information obtained from the relevant clinical letter and clinical notes

SUMMARY:
Management of pregnancy and risk stratification in congenital heart disease (CHD) population might be challenging especially due to physiological haemodynamic modifications that inevitably occur during pregnancy. We aim to compare the accuracy of the main published scores including CARPREG II score in prediction of maternal complications during pregnancy in CHD patients.

DETAILED DESCRIPTION:
Since the end of the 20th century, surgical and medical care progresses have significantly improved prognosis and quality of life of patients with congenital heart diseases (CHD). Currently, women with CHD expect to experience a "normal" life and express a strong maternity desire.

During the last decade, several scores have been used to predict outcome of pregnancy in women with cardiovascular heart diseases. It has been suggested that the mWHO classification was more appropriate than the previous ones (e.g. Harris, Zahara and CAPREG classifications) in predicting cardiac complications in CHD. More recently, a new risk score stratification (CARPREG II) have been published to improve maternal risk stratification.

This retrospective study will include all pregnant women with CHD who were follow up in our institution from January 2007 to June 2018 until 6 months postpartum. The investigators will collect demographic and clinical data, type and complexity of CHD (Houyel and Bethesda classification), and pregnancy outcomes. Pregnancy scores will be based on information obtained from the relevant clinical letter and clinical notes. The discriminatory power of each risk scores was assessed by the area-under-the receiver-operating characteristic (ROC) curve (AUC). In order to assess the reproducibility of scores classification assigned to CHD patients, all pregnancy scores from this cohort were assessed by 3 independent observers and, thereafter, estimated Cronbach's coefficient alpha.

ELIGIBILITY:
Inclusion criteria:

- All patients with congenital heart diseases who deliver in our institution during the study period

Exclusion criteria:

- Women with acquired cardiovascular diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with congenital heart diseases who delivered at Montpellier Universityhospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-12-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Number of Cardiovascular complications | From the 20th week of gestation until 6 months post partum
  Cardiovascular complications during pregnancy until 6 months post partum

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD-PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Background] Khairy P, Ionescu-Ittu R, Mackie AS, Abrahamowicz M, Pilote L, Marelli AJ. Changing mortality in congenital heart disease. J Am Coll Cardiol. 2010 Sep 28;56(14):1149-57. doi: 10.1016/j.jacc.2010.03.085. PMID 20863956
- [Background] Harris IS. Management of pregnancy in patients with congenital heart disease. Prog Cardiovasc Dis. 2011 Jan-Feb;53(4):305-11. doi: 10.1016/j.pcad.2010.08.001. PMID 21295672
- [Background] Drenthen W, Boersma E, Balci A, Moons P, Roos-Hesselink JW, Mulder BJ, Vliegen HW, van Dijk AP, Voors AA, Yap SC, van Veldhuisen DJ, Pieper PG; ZAHARA Investigators. Predictors of pregnancy complications in women with congenital heart disease. Eur Heart J. 2010 Sep;31(17):2124-32. doi: 10.1093/eurheartj/ehq200. Epub 2010 Jun 28. PMID 20584777
- [Background] Khairy P, Ouyang DW, Fernandes SM, Lee-Parritz A, Economy KE, Landzberg MJ. Pregnancy outcomes in women with congenital heart disease. Circulation. 2006 Jan 31;113(4):517-24. doi: 10.1161/CIRCULATIONAHA.105.589655. PMID 16449731
- [Background] Regitz-Zagrosek V, Roos-Hesselink JW, Bauersachs J, Blomstrom-Lundqvist C, Cifkova R, De Bonis M, Iung B, Johnson MR, Kintscher U, Kranke P, Lang IM, Morais J, Pieper PG, Presbitero P, Price S, Rosano GMC, Seeland U, Simoncini T, Swan L, Warnes CA; ESC Scientific Document Group. 2018 ESC Guidelines for the management of cardiovascular diseases during pregnancy. Eur Heart J. 2018 Sep 7;39(34):3165-3241. doi: 10.1093/eurheartj/ehy340. No abstract available. PMID 30165544
- [Background] Fu Q, Lin J. Predictive accuracy of three clinical risk assessment systems for cardiac complications among Chinese pregnant women with congenital heart disease. Int J Gynaecol Obstet. 2016 Aug;134(2):140-4. doi: 10.1016/j.ijgo.2016.02.010. Epub 2016 Apr 22. PMID 27177511
- [Background] Pijuan-Domenech A, Galian L, Goya M, Casellas M, Merced C, Ferreira-Gonzalez I, Marsal-Mora JR, Dos-Subira L, Subirana-Domenech MT, Pedrosa V, Baro-Marine F, Manrique S, Casaldaliga-Ferrer J, Tornos P, Cabero L, Garcia-Dorado D. Cardiac complications during pregnancy are better predicted with the modified WHO risk score. Int J Cardiol. 2015 Sep 15;195:149-54. doi: 10.1016/j.ijcard.2015.05.076. Epub 2015 May 15. PMID 26043149
- [Background] Cianfarani F, Masse D, Vallat G, Cano N, Guimars C, Glezer D. [The role of Regional Penitentiary Medico-Psychological Centers in the French system of aid to mental patients]. Acta Med Leg Soc (Liege). 1986;36(2):191-8. No abstract available. French. PMID 2979363
- [Derived] Bredy C, Deville F, Huguet H, Picot MC, De La Villeon G, Abassi H, Avesani M, Begue L, Burlet G, Boulot P, Fuchs F, Amedro P. Which risk score best predicts cardiovascular outcome in pregnant women with congenital heart disease? Eur Heart J Qual Care Clin Outcomes. 2023 Feb 28;9(2):177-183. doi: 10.1093/ehjqcco/qcac019. PMID 35472215